CLINICAL TRIAL: NCT01326234
Title: Further Development and Testing of an Interactive Computer-Based Program to Facilitate Readiness and Motivation for Smoking Cessation
Brief Title: Computer-Based Program to Facilitate Readiness and Motivation for Smoking Cessation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to staff changes the study never started.
Sponsor: University of Oklahoma (Other)
Responsible Party: Principal Investigator, Stephen Gillaspy, Associate Professor, University of Oklahoma
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1694
Record Dates: First submitted 2011-03-08; First posted 2011-03-30 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Smoking
Keywords: Smoking; Motivation; Cessation
MeSH Terms: conditions — Smoking | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Personalized Feedback (Active Comparator): The interactive program will provide assessment and personalized feedback on the participants' level of nicotine dependence, daily cigarette consumption, money spent on cigarettes, behavioral consequences of smoking, individual medical consequences of smoking, and family members' medical consequences of secondhand smoke.
  Interventions: Behavioral: Personalized Feedback
- Treatment as Usual (Sham Comparator): Practitioners are able to provide normal care with regard to smoking; participants will complete the Treatment Fidelity Questionnaire to assess whether any smoking cessation interventions occurred.
  Interventions: Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: Personalized Feedback — The interactive program will provide assessment and personalized feedback on the participants' level of nicotine dependence, daily cigarette consumption, money spent on cigarettes, behavioral consequences of smoking, individual medical consequences of smoking, and family members' medical consequences of secondhand smoke.
  Arms: Personalized Feedback
Behavioral: Treatment as Usual — Practitioners are able to provide normal care with regard to smoking; participants will complete the Treatment Fidelity Questionnaire to assess whether any smoking cessation interventions occurred
  Arms: Treatment as Usual

SUMMARY:
The current study seeks to use a computer-based program to target parents of children who smoke. Parents will be randomly assigned to either receive personalized feedback about their smoking behaviors or not. One month after gathering their baseline information, all participants will be asked to complete follow-up questionnaires online assessing their smoking behaviors.

DETAILED DESCRIPTION:
Tobacco use is widely recognized as the most preventable cause of cancer in the United States. Furthermore, tobacco use is responsible for 30% of all cancer-related deaths in the United States. Although practice guidelines recommend that clinicians address tobacco use during all outpatient clinic visits, the realities of the clinic setting make this difficult for overworked and overstretched clinical personnel. A computer-based intervention may enhance patient care by decreasing this burden and priming patients and families for a discussion about smoking cessation with their physician. Previous research has demonstrated the feasibility of developing and implementing an interactive computer-based program to facilitate smoking cessation in the outpatient clinic setting. The program can be self-administered, presents minimal burden to existing staff, and meets the Public Health Service practice guidelines. Furthermore, this intervention was found to be effective at increasing readiness to change in parental smoking behavior. The overall objective of this proposal is to further develop the program and test this interactive computer-based program to facilitate motivation and readiness to cease tobacco use and engage in parental smoking cessation services. The current computer program focuses on the assessment of the participant's smoking behavior and the delivery of personalized feedback regarding their smoking behavior. Modifications to the new program will include the removal of the carbon monoxide testing, inclusion of all baseline and follow-up assessment into the computer-based program (creating a single, stand-alone package that further reduces staff burden), and the inclusion of a link directly to the Oklahoma Tobacco Settlement Endowment Trust "click to call" option (allowing patients to immediately self-refer for cessation support). Parents of children presenting to a general pediatric outpatient clinic, who self-report as current smokers, will be recruited for a randomized controlled trial to assess the effectiveness of the revised computer-based program. It is proposed that exposure to this brief intervention will result in increasing smokers' readiness to cease tobacco use and engage in smoking cessation services. The successful completion of the proposed project will result in the development of a smoking cessation intervention that can be easily and consistently delivered, in a host of different settings, with little burden to existing staff. The successful development of such an intervention directly relates to the OTRC Mission and Goals and specifically fits with two of the OTRC's primary research areas: prevention and cessation of tobacco use and tobacco-related health disparities in Oklahoma's diverse populations and reduction of secondhand smoke exposure.

ELIGIBILITY:
Inclusion Criteria:

1. the parent or caregiver reports active cigarette use
2. the parent or caregiver speaks English as their primary language

Exclusion Criteria:

1. the parent or caregiver is actively attempting smoking cessation
2. the parent or caregiver reads below the 8th grade level
3. the parent or caregiver does not have email or web access

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-06; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Stage of Change | Baseline, 1- Mo Follow-up
  The Stages of Change Algorithm (SCA; DiClemente et al., 1991) will be used to categorize participants' individual stage of change in regards to smoking cessation. Participants will be asked, "Are you thinking of quitting smoking?" and then placed into one of the following stages: (1) Precontemplation, "No, I am not seriously considering quitting within the next 6 months"; (2) Contemplation, "Yes, I am seriously considering quitting within the next 6 months"; or (3) Preparation, "Yes, I am seriously planning to quit within the next 30 days."

SECONDARY OUTCOMES:
Readiness to Quit | Baseline, 1-Mo Follow-up
  The Contemplation Ladder (CL; Biener & Abrams, 1991) is a one-item instrument that provides a continuous measure of an individual's readiness to consider smoking cessation. Participants view a ladder with rungs and text ranging from 0 "No thought of quitting," to 5 "Think I should quit but am not ready," to 10 "Taking action to quit (e.g., cutting down, enrolling in a program).
Personal Importance, Confidence, and Motivation to Stop Smoking | Baseline; 1-Mo Follow-up
  Participant perception of importance, confidence, and motivation to cease tobacco use will each be measured by an 11-point rating scale, ranging from 0 (not at all) to 10 (very). Based on the stages of change model of behavior change and motivational interviewing, these three constructs are considered instrumental in assessing behavior change. The proposed format for assessing these key constructs is consistent with the typical assessment strategy used while conducting motivational interviewing (Miller & Rollnick, 2002).
Quit Behaviors | Baseline; 1-Mo follow-up
  At baseline, all participants will be asked whether they have: (1)previously quit smoking; (2)previously engaged in a quit attempt; (3) methods used to quit smoking; and (4) the length of any previous cessation periods. Additionally, during the follow-up participants will be asked whether they done any of the following since completing the program: (1) quit smoking; (2) engaged in a quit attempt; and (3) methods used to quit smoking; and (4) the length of the current smoking cessation period.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen R Gillaspy, PhD, Principal Investigator — University of Oklahoma